CLINICAL TRIAL: NCT07140757
Title: Radiofrequency Ablation for Management of Benign/Indeterminate Thyroid Nodules and Low Risk Papillary Thyroid Cancers
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-0083; NCI-2025-06179 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2025-08-22; First posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Low Risk; Papillary Thyroid Cancer; Radiofrequency Ablation
MeSH Terms: conditions — Thyroid Cancer, Papillary | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — This questionnaire includes twenty-four questions covering patients complaints ranging from 0 to 4. Patients will be asked about the presence and severity of each item currently on the medical appointment.

SUMMARY:
To track the outcomes of patients who have been treated with RFA and its long-term effectiveness, and to learn more about the quality of life of patients who have received RFA in this study.

DETAILED DESCRIPTION:
Primary Objectives

• To evaluate thyroid nodule volume changes over time in participants undergoing RFA as part of clinical care

Secondary Objectives

* To establish the health-related quality of life among participants undergoing with ultrasound guided RFA.
* To evaluate the sonographic features of thyroid nodules over time following ultrasound guided RFA.
* To assess adverse events rates following ultrasound guided RFA.

ELIGIBILITY:
Eligibility Criteria

1. Participants scheduled to undergo ultrasound-guided RFA for the following conditions: benign thyroid nodules, indeterminate thyroid nodules, low-risk DTC, and recurrent PTC
2. Participant is over 18 years and is either not a surgical candidate or has declined surgery.
3. Capable and willing to provide written informed consent
4. Participant has one of the following diagnoses:

   * Biopsy-proven benign thyroid nodules causing compressive and/or cosmetic symptoms who are requesting treatment,
   * Biopsy-proven indeterminate nodules (AUS or follicular neoplasm)
   * Papillary thyroid carcinoma (PTC) without metastasis
   * Locally recurrent thyroid cancer (< 2 cm).

Exclusion Criteria

1. Participants meeting any of the following criteria will be excluded:
2. Participants considered unsuitable for RFA by the treating physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MD Anderson Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2026-02-04 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Health- related Quality of Life Questionnaires | Through study completion; an average of 1 year
  This questionnaire includes twenty-four questions covering patients complaints ranging from 0 to 4. Patients will be asked about the presence and severity of each item currently on the medical appointment.

CONTACTS AND LOCATIONS:
Overall Officials: Victoria E Banuchi, MD, Study Director — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org